CLINICAL TRIAL: NCT01492361
Title: Evaluation of the Effect of AMR101 on Cardiovascular Health and Mortality in Hypertriglyceridemic Patients With Cardiovascular Disease or at High Risk for Cardiovascular Disease: REDUCE-IT (Reduction of Cardiovascular Events With EPA - Intervention Trial)
Brief Title: A Study of AMR101 to Evaluate Its Ability to Reduce Cardiovascular Events in High-Risk Patients With Hypertriglyceridemia and on Statin
Acronym: REDUCE-IT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amarin Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AMR-01-01-0019
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Results first posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Diseases
Keywords: Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Acute Coronary Syndrome; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Angina Pectoris; Chest Pain; Anticholesteremic Agents; Hypolipidemic Agents; Lipid Regulating Agents; Hypertriglyceridemia; Omega-3 Fatty Acids; Statin; Triglycerides; EPA; Docosahexaenoic Acid; Fish; Fatty acids; Fibrates; Niacin; Lipids; Lipoprotein; Atorvastatin; Lovaza; Simvastatin; Lovastatin; Pravastatin; Fluvastatin; Rosuvastatin; Trilipix; Vytorin; Simcor; Ezetimibe; Zetia; Ethyl-EPA; Ethyl Icosapentate; Crestor; Zocor; Lipitor; LDL; HDL; Cholesterol; Dyslipidemia; AMR101; Cardiovascular Disease, Unspecified; VASCEPA; Icosapent Ethyl
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Acute Coronary Syndrome; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Angina Pectoris; Chest Pain; Hypertriglyceridemia; Dyslipidemias | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AMR101 (Experimental): AMR101 (icosapent ethyl) + statin therapy, daily
  Interventions: Drug: AMR101; Drug: Statin therapy
- Placebo (Placebo Comparator): Placebo + statin therapy, daily
  Interventions: Drug: Placebo; Drug: Statin therapy

INTERVENTIONS:
Drug: AMR101 — Parallel Assignment
  Other Names: VASCEPA® (icosapent ethyl)
  Arms: AMR101
Drug: Placebo — Parallel Assignment
  Other Names: matching placebo
  Arms: Placebo
Drug: Statin therapy — Stable statin therapy (± ezetimibe) for at least 28 days before lipid qualification measurement (LDL-C >40 mg/dL and ≤100 mg/dL)

SUMMARY:
AMR101 (icosapent ethyl [ethyl-EPA]) is a highly purified ethyl ester of eicosapentaenoic acid (EPA) developed by Amarin Pharma Inc. for the treatment of cardiovascular disease in statin-treated patients with hypertriglyceridemia. The purpose of this study was to evaluate whether this drug, combined with a statin therapy, will be superior to the statin therapy alone, when used as a prevention in reducing long-term cardiovascular events in high-risk patients with mixed dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant or sterile women ages 45 and older
* Hypertriglyceridemia
* On statin therapy for at least four weeks
* Either having established cardiovascular disease or at high risk for cardiovascular disease

Exclusion Criteria:

* Severe heart failure
* Any life-threatening disease other than cardiovascular disease
* Active severe liver disease
* Hemoglobin A1c >10.0%
* Poorly controlled hypertension
* Planned coronary intervention (such as stent placement or heart bypass) or any non-cardiac major surgical procedure
* Known familial lipoprotein lipase deficiency (Fredrickson Type I), apolipoprotein C-II deficiency, or familial dysbetalipoproteinemia (Fredrickson Type III)
* Known hypersensitivity to the study product, fish and/or shellfish, or placebo
* History of acute or chronic pancreatitis
* Patients are excluded if using the following medications:

  * PCSK9 inhibitors
  * niacin >200 mg/day or fibrates;
  * any omega-3 fatty acid medications ;
  * dietary supplements containing omega-3 fatty acids (e.g., flaxseed oil, fish oil, krill oil, or algal oil);
  * bile acid sequestrants

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8179 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak L. Bhatt, MD, MPH, Principal Investigator — Brigham and Women's Hospital, 75 Francis Street, Boston
Locations (314):
- United States (157):
  - Amarin Investigational Site, Birmingham, Alabama
  - Amarin Investigational Site, Huntsville, Alabama
  - Amarin Investigational Site, Mobile, Alabama
  - Amarin Investigational Site, Muscle Shoals, Alabama
  - Amarin Investigational Site, Mesa, Arizona
  - Amarin Investigational Site, Phoenix, Arizona
  - Amarin Investigational Site, Tucson, Arizona
  - Amarin Investigational Site, Little Rock, Arkansas
  - Amarin Investigational Site, Beverly Hills, California
  - Amarin Investigational Site, Chino, California
  - Amarin Investigational Site, Concord, California
  - Amarin Investigational Site, El Cajon, California
  - Amarin Investigational Site, Encino, California
  - Amarin Investigational Site, Fair Oaks, California
  - Amarin Investigational Site, Hawaiian Gardens, California
  - Amarin Investigational Site, Lancaster, California
  - Amarin Investigational Site, Lincoln, California
  - Amarin Investigational Site, Los Angeles, California
  - Amarin Investigational Site, National City, California
  - Amarin Investigational Site, Orange, California
  - Amarin Investigational Site, Paramount, California
  - Amarin Investigational Site, Roseville, California
  - Amarin Investigational Site, San Diego, California
  - Amarin Investigational Site, Torrance, California
  - Amarin Investigational Site, Ventura, California
  - Amarin Investigational Site, Walnut Creek, California
  - Amarin Investigational Site, Aurora, Colorado
  - Amarin Investigational Site, Colorado Springs, Colorado
  - Amarin Investigational Site, Golden, Colorado
  - Amarin Investigational Site, Guilford, Connecticut
  - Amarin Investigational Site, Hartford, Connecticut
  - Amarin Investigational Site, Newark, Delaware
  - Amarin Investigational Site, Wilmington, Delaware
  - Amarin Investigational Site, Washington D.C., District of Columbia
  - Amarin Investigational Site, Boynton Beach, Florida
  - Amarin Investigational Site, Bradenton, Florida
  - Amarin Investigational Site, Clearwater, Florida
  - Amarin Investigational Site, Edgewater, Florida
  - Amarin Investigational Site, Fleming Island, Florida
  - Amarin Investigational Site, Fort Lauderdale, Florida
  - Amarin Investigational Site, Inverness, Florida
  - Amarin Investigational Site, Jacksonville, Florida
  - Amarin Investigational Site, Miami, Florida
  - Amarin Investigational Site, Miami Beach, Florida
  - Amarin Investigational Site, Miami Lakes, Florida
  - Amarin Investigational Site, Ocala, Florida
  - Amarin Investigational Site, Orlando, Florida
  - Amarin Investigational Site, Pembroke Pines, Florida
  - Amarin Investigational Site, Plantation, Florida
  - Amarin Investigational Site, Safety Harbor, Florida
  - Amarin Investigational Site, Sarasota, Florida
  - Amarin Investigational Site, St. Petersburg, Florida
  - Amarin Investigational Site, Vero Beach, Florida
  - Amarin Investigational Site, West Palm Beach, Florida
  - Amarin Investigational Site, Conyers, Georgia
  - Amarin Investigational Site, Covington, Georgia
  - Amarin Investigational Site, Cumming, Georgia
  - Amarin Investigational Site, Roswell, Georgia
  - Amarin Investigational Site, Honolulu, Hawaii
  - Amarin Investigational Site, Addison, Illinois
  - Amarin Investigational Site, Chicago, Illinois
  - Amarin Investigational Site, Norman, Illinois
  - Amarin Investigational Site, North Chicago, Illinois
  - Amarin Investigational Site, Peoria, Illinois
  - Amarin Investigational Site, Winfield, Illinois
  - Amarin Investigational Site, Evansville, Indiana
  - Amarin Investigational Site, Iowa City, Iowa
  - Amarin Investigational Site, Wichita, Kansas
  - Amarin Investigational Site, Louisville, Kentucky
  - Amarin Investigational Site, Alexandria, Louisiana
  - Amarin Investigational Site, Eunice, Louisiana
  - Amarin Investigational Site, Marrero, Louisiana
  - Amarin Investigational Site, Auburn, Maine
  - Amarin Investigational Site, Baltimore, Maryland
  - Amarin Investigational Site, Lutherville, Maryland
  - Amarin Investigational Site, Takoma Park, Maryland
  - Amarin Investigational Site, Boston, Massachusetts
  - Amarin Investigational Site, Fall River, Massachusetts
  - Amarin Investigational Site, Lansing, Michigan
  - Amarin Investigational Site, Marquette, Michigan
  - Amarin Investigational Site, Troy, Michigan
  - Amarin Investigational Site, Saint Cloud, Minnesota
  - Amarin Investigational Site, Biloxi, Mississippi
  - Amarin Investigational Site, Tupelo, Mississippi
  - Amarin Investigational Site, Chesterfield, Missouri
  - Amarin Investigational Site, City of Saint Peters, Missouri
  - Amarin Investigational Site, Florissant, Missouri
  - Amarin Investigational Site, Jefferson City, Missouri
  - Amarin Investigational Site, Kansas City, Missouri
  - Amarin Investigational Site, St Louis, Missouri
  - Amarin Investigational Site, Hastings, Nebraska
  - Amarin Investigational Site, Omaha, Nebraska
  - Amarin Investigational Site, Henderson, Nevada
  - Amarin Investigational Site, Las Vegas, Nevada
  - Amarin Investigational Site, Ocean City, New Jersey
  - Amarin Investigational Site, Albuquerque, New Mexico
  - Amarin Investigational Site, Albany, New York
  - Amarin Investigational Site, Brooklyn, New York
  - Amarin Investigational Site, Great Neck, New York
  - Amarin Investigational Site, Liverpool, New York
  - Amarin Investigational Site, New York, New York
  - Amarin Investigational Site, North Massapequa, New York
  - Amarin Investigational Site, Smithtown, New York
  - Amarin Investigational Site, Vestal, New York
  - Amarin Investigational Site, West Seneca, New York
  - Amarin Investigational Site, Charlotte, North Carolina
  - Amarin Investigational Site, Durham, North Carolina
  - Amarin Investigational Site, Gastonia, North Carolina
  - Amarin Investigational Site, Kernersville, North Carolina
  - Amarin Investigational Site, Raleigh, North Carolina
  - Amarin Investigational Site, Winston-Salem, North Carolina
  - Amarin Investigational Site, Fargo, North Dakota
  - Amarin Investigational Site, Cincinnati, Ohio
  - Amarin Investigational Site, Dayton, Ohio
  - Amarin Investigational Site, Lorain, Ohio
  - Amarin Investigational Site, Sandusky, Ohio
  - Amarin Investigational Site, Tulsa, Oklahoma
  - Amarin Investigational Site, Bend, Oregon
  - Amarin Investigational Site, Portland, Oregon
  - Amarin Investigational Site, Beaver, Pennsylvania
  - Amarin Investigational Site, Doylestown, Pennsylvania
  - Amarin Investigational Site, Jersey Shore, Pennsylvania
  - Amarin Investigational Site, Newport, Pennsylvania
  - Amarin Investigational Site, Philadelphia, Pennsylvania
  - Amarin Investigational Site, Phoenixville, Pennsylvania
  - Amarin Investigational Site, Sellersville, Pennsylvania
  - Amarin Investigational Site, Tipton, Pennsylvania
  - Amarin Investigational Site, Wyomissing, Pennsylvania
  - Amarin Investigational Site, Yardley, Pennsylvania
  - Amarin Investigational Site, Lancaster, South Carolina
  - Amarin Investigational Site, Simpsonville, South Carolina
  - Amarin Investigational Site, Rapid City, South Dakota
  - Amarin Investigational Site, Bristol, Tennessee
  - Amarin Investigational Site, Columbia, Tennessee
  - Amarin Investigational Site, Germantown, Tennessee
  - Amarin Investigational Site, Jackson, Tennessee
  - Amarin Investigational Site, Knoxville, Tennessee
  - Amarin Investigational Site, Smyrna, Tennessee
  - Amarin Investigational Site, Austin, Texas
  - Amarin Investigational Site, Beaumont, Texas
  - Amarin Investigational Site, Carrollton, Texas
  - Amarin Investigational Site, Dallas, Texas
  - Amarin Investigational Site, Houston, Texas
  - Amarin Investigational Site, Hurst, Texas
  - Amarin Investigational Site, New Braunfels, Texas
  - Amarin Investigational Site, Plano, Texas
  - Amarin Investigational Site, San Antonio, Texas
  - Amarin Investigational Site, Splendora, Texas
  - Amarin Investigational Site, Tomball, Texas
  - Amarin Investigational Site, West Jordan, Utah
  - Amarin Investigational Site, Falls Church, Virginia
  - Amarin Investigational Site, Manassas, Virginia
  - Amarin Investigational Site, Midlothian, Virginia
  - Amarin Investigational Site, Newport News, Virginia
  - Amarin Investigational Site, Burien, Washington
  - Amarin Investigational Site, Tacoma, Washington
  - Amarin Investigational Site, Huntington, West Virginia
- Australia (15):
  - Amarin Investigational Site, Camperdown, New South Wales
  - Amarin Investigational Site, Lismore, New South Wales
  - Amarin Investigational Site, Brisbane, Queensland
  - Amarin Investigational Site, Chermside, Queensland
  - Amarin Investigational Site, Bedford Park, South Australia
  - Amarin Investigational Site, Launceston, Tasmania
  - Amarin Investigational Site, Fitzroy, Victoria
  - Amarin Investigational Site, Geelong, Victoria
  - Amarin Investigational Site, Heidelberg Heights, Victoria
  - Amarin Investigational Site, Melbourne, Victoria
  - Amarin Investigational Site, Fremantle, Western Australia
  - Amarin Investigational Site, Joondalup, Western Australia
  - Amarin Investigational Site, Murdoch, Western Australia
  - Amarin Investigational Site, Nedlands, Western Australia
  - Amarin Investigational Site, Perth, Western Australia
- Canada (14):
  - Amarin Investigational Site, Edmonton, Alberta
  - Amarin Investigational Site, Coquitlam, British Columbia
  - Amarin Investigational Site, Vancouver, British Columbia
  - Amarin Investigational Site, Brampton, Ontario
  - Amarin Investigational Site, Collingwood, Ontario
  - Amarin Investigational Site, Corunna, Ontario
  - Amarin Investigational Site, Newmarket, Ontario
  - Amarin Investigational Site, Sarnia, Ontario
  - Amarin Investigational Site, Strathroy, Ontario
  - Amarin Investigational Site, Laval, Quebec
  - Amarin Investigational Site, Montreal, Quebec
  - Amarin Investigational Site, Saint-Charles-Borromée, Quebec
  - Amarin Investigational Site, Sherbrooke, Quebec
  - Amarin Investigational Site, Québec
- India (12):
  - Amarin Investigational Site, Hyderabad, Andhra Pradesh
  - Amarin Investigational Site, Secunderabad, Andhra Pradesh
  - Amarin Investigational Site, Visakhapatnam, Andhra Pradesh
  - Amarin Investigational Site, Bangalore, Karnataka
  - Amarin Investigational Site, Mysore, Karnataka
  - Amarin Investigational Site, Kottayam, Kerala
  - Amarin Investigational Site, Mumbai, Maharashtra
  - Amarin Investigational Site, Nashik, Maharashtra
  - Amarin Investigational Site, Pune, Maharashtra
  - Amarin Investigational Site, New Delhi, National Capital Territory of Delhi
  - Amarin Investigational Site, Chennai, Tamil Nadu
  - Amarin Investigational Site, Coimbatore, Tamil Nadu
- Netherlands (32):
  - Amarin Investigational Site, Almelo
  - Amarin Investigational Site, Amersfoort
  - Amarin Investigational Site, Blaricum
  - Amarin Investigational Site, Capelle aan den IJssel
  - Amarin Investigational Site, Den Helder
  - Amarin Investigational Site, Deventer
  - Amarin Investigational Site, Ede
  - Amarin Investigational Site, Eindhoven
  - Amarin Investigational Site, Enschede
  - Amarin Investigational Site, Goes
  - Amarin Investigational Site, Gorinchem
  - Amarin Investigational Site, Gouda
  - Amarin Investigational Site, Groningen
  - Amarin Investigational Site, Haarlem
  - Amarin Investigational Site, Harderwijk
  - Amarin Investigational Site, Heerenveen
  - Amarin Investigational Site, Heerlen
  - Amarin Investigational Site, Hoofddorp
  - Amarin Investigational Site, Leeuwarden
  - Amarin Investigational Site, Leiderdorp
  - Amarin Investigational Site, Nijmegen
  - Amarin Investigational Site, Roosendaal
  - Amarin Investigational Site, Rotterdam
  - Amarin Investigational Site, s'Hertogenbosch
  - Amarin Investigational Site, Schiedam
  - Amarin Investigational Site, Sneek
  - Amarin Investigational Site, The Hague
  - Amarin Investigational Site, Tilburg
  - Amarin Investigational Site, Uden
  - Amarin Investigational Site, Veldhoven
  - Amarin Investigational Site, Zoetermeer
  - Amarin Investigational Site, Zutphen
- New Zealand (10):
  - Amarin Investigational Site, Takapuna, Auckland
  - Amarin Investigational Site, Christchurch
  - Amarin Investigational Site, Dunedin
  - Amarin Investigational Site, Hamilton
  - Amarin Investigational Site, Hastings
  - Amarin Investigational Site, Nelson
  - Amarin Investigational Site, New Plymouth
  - Amarin Investigational Site, Takapuna Auckland
  - Amarin Investigational Site, Tauranga
  - Amarin Investigational Site, Whangarei
- Poland (10):
  - Amarin Investigational Site, Bialystok
  - Amarin Investigational Site, Katowice
  - Amarin Investigational Site, Krakow
  - Amarin Investigational Site, Mikolów
  - Amarin Investigational Site, Skierniewice
  - Amarin Investigational Site, Tarnów
  - Amarin Investigational Site, Warsaw
  - Amarin Investigational Site, Warszawska
  - Amarin Investigational Site, Wroclaw
  - Amarin Investigational Site, Zgierz
- Romania (12):
  - Amarin Investigational Site, Argeş
  - Amarin Investigational Site, Brăila
  - Amarin Investigational Site, Bucharest
  - Amarin Investigational Site, Cluj-Napoca
  - Amarin Investigational Site, Constanța
  - Amarin Investigational Site, Craiova, Dolj
  - Amarin Investigational Site, Iași
  - Amarin Investigational Site, Maramureş
  - Amarin Investigational Site, Mureş
  - Amarin Investigational Site, Sibiu
  - Amarin Investigational Site, Târgu Mureş
  - Amarin Investigational Site, Timișoara
- Russia (17):
  - Amarin Investigational Site, Arkhangelsk
  - Amarin Investigational Site, Kazan'
  - Amarin Investigational Site, Kemerovo
  - Amarin Investigational Site, Kirovsk, Leningradskaya Region
  - Amarin Investigational Site, Krasnodar
  - Amarin Investigational Site, Moscow
  - Amarin Investigational Site, Nizhny Novgorod
  - Amarin Investigational Site, Novosibirsk
  - Amarin Investigational Site, Petrozavodsk
  - Amarin Investigational Site, Saint Petersburg
  - Amarin Investigational Site, Saratov
  - Amarin Investigational Site, Sestroretsk, Saint-Petersburg
  - Amarin Investigational Site, Tomsk
  - Amarin Investigational Site, Volgograd
  - Amarin Investigational Site, Voronezh
  - Amarin Investigational Site, Yaroslavl
  - Amarin Investigational Site, Yekaterinburg
- South Africa (18):
  - Amarin Investigational Site, Bloemfontein, Freestate
  - Amarin Investigational Site, Benoni, Gauteng
  - Amarin Investigational Site, Pretoria, Gauteng
  - Amarin Investigational Site, Soweto, Gauteng
  - Amarin Investigational Site, Witbank, Gauteng
  - Amarin Investigational Site, Durban, KwaZulu-Natal
  - Amarin Investigational Site, Newlands, KwaZulu-Natal
  - Amarin Investigational Site, Bellville, Western Cape
  - Amarin Investigational Site, Cape Town, Western Cape
  - Amarin Investigational Site, Durbanville, Western Cape
  - Amarin Investigational Site, Goodwood, Western Cape
  - Amarin Investigational Site, Kraaifontein, Western Cape
  - Amarin Investigational Site, Paarl, Western Cape
  - Amarin Investigational Site, Panorama, Western Cape
  - Amarin Investigational Site, Parow, Western Cape
  - Amarin Investigational Site, Pinelands, Western Cape
  - Amarin Investigational Site, Somerset West, Western Cape
  - Amarin Investigational Site, Worcester, Western Cape
- Ukraine (17):
  - Amarin Investigational Site, Lutsk, Volyn Oblast
  - Amarin Investigational Site, Cherkasy
  - Amarin Investigational Site, Chernivtsi
  - Amarin Investigational Site, Dnipropetrovsk
  - Amarin Investigational Site, Donetsk
  - Amarin Investigational Site, Ivano-Frankivsk
  - Amarin Investigational Site, Kharkiv
  - Amarin Investigational Site, Kyiv
  - Amarin Investigational Site, Luhansk
  - Amarin Investigational Site, Lutsk
  - Amarin Investigational Site, Lviv
  - Amarin Investigational Site, Odesa
  - Amarin Investigational Site, Poltava
  - Amarin Investigational Site, Ternopil
  - Amarin Investigational Site, Uzhhorod
  - Amarin Investigational Site, Vinnytsia
  - Amarin Investigational Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhatt DL, Steg PG, Brinton EA, Jacobson TA, Miller M, Tardif JC, Ketchum SB, Doyle RT Jr, Murphy SA, Soni PN, Braeckman RA, Juliano RA, Ballantyne CM; REDUCE-IT Investigators. Rationale and design of REDUCE-IT: Reduction of Cardiovascular Events with Icosapent Ethyl-Intervention Trial. Clin Cardiol. 2017 Mar;40(3):138-148. doi: 10.1002/clc.22692. Epub 2017 Mar 15. PMID 28294373
- [Result] Bhatt DL, Steg PG, Miller M, Brinton EA, Jacobson TA, Ketchum SB, Doyle RT Jr, Juliano RA, Jiao L, Granowitz C, Tardif JC, Ballantyne CM; REDUCE-IT Investigators. Cardiovascular Risk Reduction with Icosapent Ethyl for Hypertriglyceridemia. N Engl J Med. 2019 Jan 3;380(1):11-22. doi: 10.1056/NEJMoa1812792. Epub 2018 Nov 10. PMID 30415628
- [Result] Bhatt DL, Steg PG, Miller M, Brinton EA, Jacobson TA, Ketchum SB, Doyle RT Jr, Juliano RA, Jiao L, Granowitz C, Tardif JC, Gregson J, Pocock SJ, Ballantyne CM; REDUCE-IT Investigators. Effects of Icosapent Ethyl on Total Ischemic Events: From REDUCE-IT. J Am Coll Cardiol. 2019 Jun 11;73(22):2791-2802. doi: 10.1016/j.jacc.2019.02.032. Epub 2019 Mar 18. PMID 30898607
- [Result] Bhatt DL, Miller M, Brinton EA, Jacobson TA, Steg PG, Ketchum SB, Doyle RT Jr, Juliano RA, Jiao L, Granowitz C, Tardif JC, Olshansky B, Chung MK, Gibson CM, Giugliano RP, Budoff MJ, Ballantyne CM; REDUCE-IT Investigators. REDUCE-IT USA: Results From the 3146 Patients Randomized in the United States. Circulation. 2020 Feb 4;141(5):367-375. doi: 10.1161/CIRCULATIONAHA.119.044440. Epub 2019 Nov 11. PMID 31707829
- [Result] Olshansky B, Bhatt DL, Miller M, Steg PG, Brinton EA, Jacobson TA, Ketchum SB, Doyle RT Jr, Juliano RA, Jiao L, Granowitz C, Tardif JC, Mehta C, Mukherjee R, Ballantyne CM, Chung MK; REDUCE-IT Investigators. REDUCE-IT INTERIM: accumulation of data across prespecified interim analyses to final results. Eur Heart J Cardiovasc Pharmacother. 2021 May 23;7(3):e61-e63. doi: 10.1093/ehjcvp/pvaa118. No abstract available. PMID 33010162
- [Result] Peterson BE, Bhatt DL, Steg PG, Miller M, Brinton EA, Jacobson TA, Ketchum SB, Juliano RA, Jiao L, Doyle RT Jr, Granowitz C, Gibson CM, Pinto D, Giugliano RP, Budoff MJ, Tardif JC, Verma S, Ballantyne CM; REDUCE-IT Investigators. Reduction in Revascularization With Icosapent Ethyl: Insights From REDUCE-IT Revascularization Analyses. Circulation. 2021 Jan 5;143(1):33-44. doi: 10.1161/CIRCULATIONAHA.120.050276. Epub 2020 Nov 5. PMID 33148016
- [Result] Bhatt DL, Steg PG, Miller M, Brinton EA, Jacobson TA, Jiao L, Tardif JC, Gregson J, Pocock SJ, Ballantyne CM; REDUCE-IT Investigators. Reduction in First and Total Ischemic Events With Icosapent Ethyl Across Baseline Triglyceride Tertiles. J Am Coll Cardiol. 2019 Aug 27;74(8):1159-1161. doi: 10.1016/j.jacc.2019.06.043. No abstract available. PMID 31439224
- [Result] Gaba P, Bhatt DL, Giugliano RP, Steg PG, Miller M, Brinton EA, Jacobson TA, Ketchum SB, Juliano RA, Jiao L, Doyle RT Jr, Granowitz C, Tardif JC, Ballantyne CM, Pinto DS, Budoff MJ, Gibson CM. Comparative Reductions in Investigator-Reported and Adjudicated Ischemic Events in REDUCE-IT. J Am Coll Cardiol. 2021 Oct 12;78(15):1525-1537. doi: 10.1016/j.jacc.2021.08.009. PMID 34620410
- [Result] Majithia A, Bhatt DL, Friedman AN, Miller M, Steg PG, Brinton EA, Jacobson TA, Ketchum SB, Juliano RA, Jiao L, Doyle RT Jr, Granowitz C, Budoff M, Preston Mason R, Tardif JC, Boden WE, Ballantyne CM. Benefits of Icosapent Ethyl Across the Range of Kidney Function in Patients With Established Cardiovascular Disease or Diabetes: REDUCE-IT RENAL. Circulation. 2021 Nov 30;144(22):1750-1759. doi: 10.1161/CIRCULATIONAHA.121.055560. Epub 2021 Oct 28. PMID 34706555
- [Result] Verma S, Bhatt DL, Steg PG, Miller M, Brinton EA, Jacobson TA, Dhingra NK, Ketchum SB, Juliano RA, Jiao L, Doyle RT Jr, Granowitz C, Gibson CM, Pinto D, Giugliano RP, Budoff MJ, Mason RP, Tardif JC, Ballantyne CM; REDUCE-IT Investigators. Icosapent Ethyl Reduces Ischemic Events in Patients With a History of Previous Coronary Artery Bypass Grafting: REDUCE-IT CABG. Circulation. 2021 Dec 7;144(23):1845-1855. doi: 10.1161/CIRCULATIONAHA.121.056290. Epub 2021 Oct 28. PMID 34710343
- [Result] Singh N, Bhatt DL, Miller M, Steg PG, Brinton EA, Jacobson TA, Jiao L, Tardif JC, Mason RP, Ballantyne CM; REDUCE-IT Investigators. Consistency of Benefit of Icosapent Ethyl by Background Statin Type in REDUCE-IT. J Am Coll Cardiol. 2022 Jan 18;79(2):220-222. doi: 10.1016/j.jacc.2021.11.005. No abstract available. PMID 35027114
- [Derived] Gurevitz C, Bhatt DL, Giugliano RP, Steg PG, Miller M, Brinton EA, Jacobson TA, Ketchum SB, Lira Pineda A, Doyle RT Jr, Giugliano G, Mason RP, Tardif JC, Martens FMAC, Ballantyne CM, Budoff MJ, Gibson CM. Benefit of Icosapent Ethyl Across Types and Sizes of Myocardial Infarction in REDUCE-IT. Eur J Prev Cardiol. 2025 Sep 22:zwaf602. doi: 10.1093/eurjpc/zwaf602. Online ahead of print. PMID 40982548
- [Derived] Aggarwal R, Bhatt DL, Steg PG, Miller M, Brinton EA, Dunbar RL, Ketchum SB, Tardif JC, Martens FMAC, Ballantyne CM, Szarek M, Mason RP; REDUCE-IT Investigators. Cardiovascular Outcomes With Icosapent Ethyl by Baseline Low-Density Lipoprotein Cholesterol: A Secondary Analysis of the REDUCE-IT Randomized Trial. J Am Heart Assoc. 2025 Mar 4;14(5):e038656. doi: 10.1161/JAHA.124.038656. Epub 2025 Feb 19. PMID 39968782
- [Derived] Weintraub WS, Bhatt DL, Zhang Z, Dolman S, Boden WE, Bress AP, Bellows BK, Derington CG, Philip S, Steg G, Miller M, Brinton EA, Jacobson TA, Tardif JC, Ballantyne CM, Kolm P. Cost-Effectiveness of Icosapent Ethyl in REDUCE-IT USA: Results From Patients Randomized in the United States. J Am Heart Assoc. 2024 Jan 2;13(1):e032413. doi: 10.1161/JAHA.123.032413. Epub 2023 Dec 29. PMID 38156550
- [Derived] Miller M, Bhatt DL, Brinton EA, Jacobson TA, Steg PG, Pineda AL, Ketchum SB, Doyle RT Jr, Tardif JC, Ballantyne CM. Effectiveness of icosapent ethyl on first and total cardiovascular events in patients with metabolic syndrome, but without diabetes: REDUCE-IT MetSyn. Eur Heart J Open. 2023 Nov 12;3(6):oead114. doi: 10.1093/ehjopen/oead114. eCollection 2023 Nov. PMID 38035037
- [Derived] Olshansky B, Bhatt DL, Miller M, Steg PG, Brinton EA, Jacobson TA, Ketchum SB, Doyle RT Jr, Juliano RA, Jiao L, Kowey PR, Reiffel JA, Tardif JC, Ballantyne CM, Chung MK; REDUCE-IT Investigators. Cardiovascular Benefits of Icosapent Ethyl in Patients With and Without Atrial Fibrillation in REDUCE-IT. J Am Heart Assoc. 2023 Mar 7;12(5):e026756. doi: 10.1161/JAHA.121.026756. Epub 2023 Feb 21. PMID 36802845
- [Derived] Ridker PM, Rifai N, MacFadyen J, Glynn RJ, Jiao L, Steg PG, Miller M, Brinton EA, Jacobson TA, Tardif JC, Ballantyne CM, Mason RP, Bhatt DL. Effects of Randomized Treatment With Icosapent Ethyl and a Mineral Oil Comparator on Interleukin-1beta, Interleukin-6, C-Reactive Protein, Oxidized Low-Density Lipoprotein Cholesterol, Homocysteine, Lipoprotein(a), and Lipoprotein-Associated Phospholipase A2: A REDUCE-IT Biomarker Substudy. Circulation. 2022 Aug 2;146(5):372-379. doi: 10.1161/CIRCULATIONAHA.122.059410. Epub 2022 Jun 28. PMID 35762321
- [Derived] Gaba P, Bhatt DL, Steg PG, Miller M, Brinton EA, Jacobson TA, Ketchum SB, Juliano RA, Jiao L, Doyle RT Jr, Granowitz C, Tardif JC, Giugliano RP, Martens FMAC, Gibson CM, Ballantyne CM; REDUCE-IT Investigators. Prevention of Cardiovascular Events and Mortality With Icosapent Ethyl in Patients With Prior Myocardial Infarction. J Am Coll Cardiol. 2022 May 3;79(17):1660-1671. doi: 10.1016/j.jacc.2022.02.035. PMID 35483753
- [Derived] Selvaraj S, Bhatt DL, Steg PG, Miller M, Brinton EA, Jacobson TA, Juliano RA, Jiao L, Tardif JC, Ballantyne CM; REDUCE-IT Investigators. Impact of Icosapent Ethyl on Cardiovascular Risk Reduction in Patients With Heart Failure in REDUCE-IT. J Am Heart Assoc. 2022 Apr 5;11(7):e024999. doi: 10.1161/JAHA.121.024999. Epub 2022 Apr 4. PMID 35377160
- [Derived] Peterson BE, Bhatt DL, Steg PG, Miller M, Brinton EA, Jacobson TA, Ketchum SB, Juliano RA, Jiao L, Doyle RT Jr, Granowitz C, Gibson CM, Pinto D, Giugliano RP, Budoff MJ, Tardif JC, Verma S, Ballantyne CM; REDUCE-IT Investigators. Treatment With Icosapent Ethyl to Reduce Ischemic Events in Patients With Prior Percutaneous Coronary Intervention: Insights From REDUCE-IT PCI. J Am Heart Assoc. 2022 Mar 15;11(6):e022937. doi: 10.1161/JAHA.121.022937. Epub 2022 Mar 9. PMID 35261279

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AMR101 | Placebo
Started | 4089 | 4090
Completed Final Visit | 3419 | 3335
Death Before Final Visit (Participants who died on trial were considered completed) | 265 | 295
Completed | 3684 | 3630
Not Completed | 405 | 460
Not completed — Withdrawal by Subject | 281 | 297
Not completed — Physician Decision | 12 | 12
Not completed — Lost to Follow-up | 6 | 13
Not completed — Other than specified above | 106 | 138

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AMR101 | Placebo | Total
Number analyzed (Participants) | 4089 | 4090 | 8179
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.0 [57.0 to 69.0] | 64.0 [57.0 to 69.0] | 64.0 [57.0 to 69.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1162 | 1195 | 2357
  Male | 2927 | 2895 | 5822
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 3691 | 3688 | 7379
  Race: Other than white | 398 | 401 | 799
  Race: Missing | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  New Zealand | 73 | 61 | 134
  Canada | 123 | 127 | 250
  Netherlands | 847 | 831 | 1678
  Romania | 109 | 93 | 202
  United States | 1548 | 1598 | 3146
  Ukraine | 397 | 439 | 836
  Poland | 195 | 164 | 359
  South Africa | 213 | 201 | 414
  Australia | 102 | 87 | 189
  India | 130 | 132 | 262
  Russia | 352 | 357 | 709
Cardiovascular Risk Stratum [Count of Participants; unit: Participants]
  Secondary-prevention cohort | 2892 | 2893 | 5785
  Primary-prevention cohort | 1197 | 1197 | 2394

OUTCOME MEASURES:

1. Primary Outcome: Composite of CV Death, Nonfatal MI (Including Silent MI), Nonfatal Stroke, Coronary Revascularization, or Unstable Angina Determined to be Caused by Myocardial Ischemia by Invasive / Non-invasive Testing and Requiring Emergent Hospitalization.
Description: The primary outcome measure was the number of patients with a first occurrence of any component of the composite of CV death, nonfatal MI (including silent MI), nonfatal stroke, coronary revascularization, or unstable angina determined to be caused by myocardial ischemia by invasive / non-invasive testing and requiring emergent hospitalization during the follow-up period.
Time Frame: Total follow-up time of up to approximately 6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | AMR101 | Placebo
Number analyzed (Participants) | 4089 | 4090
Participants | 705 | 901
Statistical Analysis 1: Comparison: AMR101 vs Placebo; Test type: Superiority; p = 0.00000001, Log Rank — The 2-sided alpha level for the primary analysis was adjusted to 0.0437 from 0.05 to account for the two interim analyses based on a group sequential design with O'Brien-Fleming boundaries generated using the Lan-DeMets alpha-spending function; Stratified by CV risk category, use of ezetimibe, and geographical region; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.68 to 0.83]

2. Secondary Outcome: Composite of CV Death, Nonfatal MI (Including Silent MI), or Nonfatal Stroke.
Description: The key secondary outcome measure was the number of patients with a first occurrence of any component of the composite of CV death, nonfatal MI (including silent MI), or nonfatal stroke during the follow-up period.
Time Frame: Total follow-up time of up to approximately 6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | AMR101 | Placebo
Number analyzed (Participants) | 4089 | 4090
Participants | 459 | 606
Statistical Analysis 1: Comparison: AMR101 vs Placebo; Test type: Superiority; p = 0.0000006, Log Rank — Prespecified secondary end points were tested in a hierarchical fashion, in the order listed here, at the final alpha level of 0.0437; Stratified by CV risk category, use of ezetimibe, and geographical region; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.65 to 0.83]

3. Secondary Outcome: Composite of CV Death or Nonfatal MI (Including Silent MI).
Description: Number of patients with a first occurrence of any component of the composite of CV death or nonfatal MI (including silent MI) during the follow-up period.
Time Frame: Total follow-up time of up to approximately 6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | AMR101 | Placebo
Number analyzed (Participants) | 4089 | 4090
Participants | 392 | 507
Statistical Analysis 1: Comparison: AMR101 vs Placebo; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Stratified by CV risk category, use of ezetimibe, and geographical region; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.66 to 0.86]

4. Secondary Outcome: Fatal or Nonfatal MI (Including Silent MI).
Description: Number of patients with a first occurrence of fatal or nonfatal MI (including silent MI) during the follow-up period.
Time Frame: Total follow-up time of up to approximately 6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | AMR101 | Placebo
Number analyzed (Participants) | 4089 | 4090
Participants | 250 | 355
Statistical Analysis 1: Comparison: AMR101 vs Placebo; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Stratified by CV risk category, use of ezetimibe, and geographical region; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.58 to 0.81]

5. Secondary Outcome: Non-elective Coronary Revascularization Represented as the Composite of Emergent or Urgent Classifications.
Description: Number of patients with a first occurrence of non-elective coronary revascularization represented as the composite of emergent or urgent classifications during the follow-up period.
Time Frame: Total follow-up time of up to approximately 6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | AMR101 | Placebo
Number analyzed (Participants) | 4089 | 4090
Participants | 216 | 321
Statistical Analysis 1: Comparison: AMR101 vs Placebo; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Stratified by CV risk category, use of ezetimibe, and geographical region; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.55 to 0.78]

6. Secondary Outcome: CV Death.
Description: Number of patients with an occurrence of CV death during the follow-up period.
Time Frame: Total follow-up time of up to approximately 6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | AMR101 | Placebo
Number analyzed (Participants) | 4089 | 4090
Participants | 174 | 213
Statistical Analysis 1: Comparison: AMR101 vs Placebo; Test type: Superiority; p = 0.0315, Log Rank — [p-value comment as in outcome 2, analysis 1]; Stratified by CV risk category, use of ezetimibe, and geographical region; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.66 to 0.98]

7. Secondary Outcome: Unstable Angina Determined to be Caused by Myocardial Ischemia by Invasive / Non-invasive Testing and Requiring Emergent Hospitalization.
Description: Number of patients with a first occurrence of unstable angina determined to be caused by myocardial ischemia by invasive / non-invasive testing and requiring emergent hospitalization during the follow-up period.
Time Frame: Total follow-up time of up to approximately 6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | AMR101 | Placebo
Number analyzed (Participants) | 4089 | 4090
Participants | 108 | 157
Statistical Analysis 1: Comparison: AMR101 vs Placebo; Test type: Superiority; p = 0.0018, Log Rank — [p-value comment as in outcome 2, analysis 1]; Stratified by CV risk category, use of ezetimibe, and geographical region; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.53 to 0.87]

8. Secondary Outcome: Fatal or Nonfatal Stroke.
Description: Number of patients with a first occurrence of fatal or nonfatal stroke during the follow-up period.
Time Frame: Total follow-up time of up to approximately 6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | AMR101 | Placebo
Number analyzed (Participants) | 4089 | 4090
Participants | 98 | 134
Statistical Analysis 1: Comparison: AMR101 vs Placebo; Test type: Superiority; p = 0.0129, Log Rank — [p-value comment as in outcome 2, analysis 1]; Stratified by CV risk category, use of ezetimibe, and geographical region; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.55 to 0.93]

9. Secondary Outcome: Total Mortality, Nonfatal MI (Including Silent MI), or Nonfatal Stroke.
Description: Number of patients with a first occurrence of any component of the composite of total mortality, nonfatal MI (including silent MI), or nonfatal stroke during the follow-up period.
Time Frame: Total follow-up time of up to approximately 6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | AMR101 | Placebo
Number analyzed (Participants) | 4089 | 4090
Participants | 549 | 690
Statistical Analysis 1: Comparison: AMR101 vs Placebo; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Stratified by CV risk category, use of ezetimibe, and geographical region; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.69 to 0.86]

10. Secondary Outcome: Total Mortality.
Description: Number of patients with an occurrence of death from any cause during the follow-up period.
Time Frame: Total follow-up time of up to approximately 6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | AMR101 | Placebo
Number analyzed (Participants) | 4089 | 4090
Participants | 274 | 310
Statistical Analysis 1: Comparison: AMR101 vs Placebo; Test type: Superiority; p = 0.0915, Log Rank — [p-value comment as in outcome 2, analysis 1]; Stratified by CV risk category, use of ezetimibe, and geographical region; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.74 to 1.02]

ADVERSE EVENTS:
Time Frame: Up to maximum duration of approximate 6 years from first dose of study treatment until end of study treatment plus 30 days post treatment.
Description: Adverse events were collected from first dose of study treatment until the completion or withdrawal from study plus 30 days post treatment.
Arm/Group | AMR101 | Placebo
All-Cause Mortality (participants affected / at risk) | 274/4089 | 310/4090
Serious Adverse Events (participants affected / at risk) | 1252/4089 | 1254/4090
Other Adverse Events (participants affected / at risk) | 3268/4089 | 3248/4090
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMR101 (N=4089) | Placebo (N=4090)
Pneumonia (Infections and infestations) | 105 | 118
Cellulitis (Infections and infestations) | 36 | 28
Sepsis (Infections and infestations) | 25 | 31
Urinary tract infection (Infections and infestations) | 25 | 22
Gastroenteritis (Infections and infestations) | 16 | 16
Erysipelas (Infections and infestations) | 13 | 3
Osteomyelitis (Infections and infestations) | 12 | 7
Septic shock (Infections and infestations) | 12 | 3
Bronchitis (Infections and infestations) | 11 | 10
Diverticulitis (Infections and infestations) | 11 | 9
Urosepsis (Infections and infestations) | 11 | 9
Appendicitis (Infections and infestations) | 9 | 6
Postoperative wound infection (Infections and infestations) | 8 | 4
Pyelonephritis (Infections and infestations) | 7 | 4
Gastroenteritis viral (Infections and infestations) | 5 | 1
Arthritis bacterial (Infections and infestations) | 4 | 2
Wound infection (Infections and infestations) | 4 | 2
Bacteraemia (Infections and infestations) | 3 | 4
Cystitis (Infections and infestations) | 3 | 3
Localised infection (Infections and infestations) | 3 | 3
Arthritis infective (Infections and infestations) | 3 | 2
Staphylococcal infection (Infections and infestations) | 3 | 2
Abscess limb (Infections and infestations) | 3 | 1
Gangrene (Infections and infestations) | 3 | 1
Intervertebral discitis (Infections and infestations) | 3 | 1
Laryngitis (Infections and infestations) | 3 | 0
Influenza (Infections and infestations) | 2 | 4
Pyelonephritis acute (Infections and infestations) | 2 | 4
Anal abscess (Infections and infestations) | 2 | 2
Herpes zoster (Infections and infestations) | 2 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 1
Liver abscess (Infections and infestations) | 2 | 1
Appendicitis perforated (Infections and infestations) | 2 | 0
Meningitis bacterial (Infections and infestations) | 2 | 0
Necrotising fasciitis (Infections and infestations) | 2 | 0
Parainfluenzae virus infection (Infections and infestations) | 2 | 0
Perirectal abscess (Infections and infestations) | 2 | 0
Pneumococcal sepsis (Infections and infestations) | 2 | 0
Pneumonia streptococcal (Infections and infestations) | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 5
Endocarditis (Infections and infestations) | 1 | 4
Viral infection (Infections and infestations) | 1 | 3
Abscess intestinal (Infections and infestations) | 1 | 2
Clostridium difficile infection (Infections and infestations) | 1 | 2
Implant site infection (Infections and infestations) | 1 | 2
Peritonitis (Infections and infestations) | 1 | 2
Pneumonia staphylococcal (Infections and infestations) | 1 | 2
Bronchitis viral (Infections and infestations) | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 1
Gastroenteritis rotavirus (Infections and infestations) | 1 | 1
Pneumonia influenzal (Infections and infestations) | 1 | 1
Pneumonia pseudomonal (Infections and infestations) | 1 | 1
Postoperative abscess (Infections and infestations) | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 1
Tracheobronchitis (Infections and infestations) | 1 | 1
Acquired immunodeficiency syndrome (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Catheter site cellulitis (Infections and infestations) | 1 | 0
Cellulitis streptococcal (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cystitis bacterial (Infections and infestations) | 1 | 0
Cystitis escherichia (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Epiglottitis (Infections and infestations) | 1 | 0
Gastrointestinal bacterial overgrowth (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Genital infection fungal (Infections and infestations) | 1 | 0
Graft infection (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 1 | 0
Incision site abscess (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Infectious colitis (Infections and infestations) | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0
Joint abscess (Infections and infestations) | 1 | 0
Keratitis bacterial (Infections and infestations) | 1 | 0
Latent tuberculosis (Infections and infestations) | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Mycobacterial infection (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pharyngolaryngeal abscess (Infections and infestations) | 1 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Shunt infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subacute endocarditis (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0
Tick-borne fever (Infections and infestations) | 1 | 0
Viral sepsis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulval cellulitis (Infections and infestations) | 1 | 0
Wound sepsis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 2
Orchitis (Infections and infestations) | 0 | 2
Rotavirus infection (Infections and infestations) | 0 | 2
Abdominal abscess (Infections and infestations) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Biliary abscess (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1
Bursitis infective (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Gas gangrene (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Listeriosis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Osteomyelitis acute (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1
Parasitic gastroenteritis (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Pyelocystitis (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1
Sepsis syndrome (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Wound abscess (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 | 26
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 8
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 6
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 14
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 9
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 9
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer male (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Extranodal marginal zone B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Iris melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian granulosa-theca cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mucoepidermoid carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian epithelial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Refractory anaemia with ringed sideroblasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Refractory cytopenia with unilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angina pectoris (Cardiac disorders) | 48 | 48
Angina unstable (Cardiac disorders) | 41 | 53
Atrial fibrillation (Cardiac disorders) | 21 | 17
Cardiac failure congestive (Cardiac disorders) | 19 | 13
Aortic valve stenosis (Cardiac disorders) | 10 | 7
Coronary artery disease (Cardiac disorders) | 9 | 16
Cardiac failure (Cardiac disorders) | 7 | 8
Acute coronary syndrome (Cardiac disorders) | 6 | 4
Myocardial infarction (Cardiac disorders) | 4 | 12
Cardiac arrest (Cardiac disorders) | 4 | 9
Myocardial ischaemia (Cardiac disorders) | 4 | 4
Cardiomyopathy (Cardiac disorders) | 4 | 2
Mitral valve incompetence (Cardiac disorders) | 4 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 3 | 3
Arrhythmia (Cardiac disorders) | 3 | 2
Palpitations (Cardiac disorders) | 3 | 1
Cardiac failure acute (Cardiac disorders) | 3 | 0
Ventricular arrhythmia (Cardiac disorders) | 3 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 3
Pericarditis (Cardiac disorders) | 2 | 3
Ventricular tachycardia (Cardiac disorders) | 2 | 1
Left ventricular failure (Cardiac disorders) | 2 | 0
Supraventricular extrasystoles (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 4
Atrial flutter (Cardiac disorders) | 1 | 3
Aortic valve incompetence (Cardiac disorders) | 1 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 2
Coronary artery stenosis (Cardiac disorders) | 1 | 2
Left ventricular dysfunction (Cardiac disorders) | 1 | 2
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cor pulmonale chronic (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Pleuropericarditis (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Ventricular parasystole (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 4
Cardiac tamponade (Cardiac disorders) | 0 | 3
Arteriospasm coronary (Cardiac disorders) | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 2
Silent myocardial infarction (Cardiac disorders) | 0 | 2
Ventricular fibrillation (Cardiac disorders) | 0 | 2
Aortic valve disease (Cardiac disorders) | 0 | 1
Aortic valve disease mixed (Cardiac disorders) | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery dissection (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Microvascular coronary artery disease (Cardiac disorders) | 0 | 1
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 26 | 20
Small intestinal obstruction (Gastrointestinal disorders) | 16 | 12
Inguinal hernia (Gastrointestinal disorders) | 11 | 8
Rectal haemorrhage (Gastrointestinal disorders) | 10 | 6
Abdominal pain (Gastrointestinal disorders) | 7 | 4
Vomiting (Gastrointestinal disorders) | 7 | 4
Constipation (Gastrointestinal disorders) | 6 | 8
Colitis (Gastrointestinal disorders) | 6 | 6
Abdominal pain upper (Gastrointestinal disorders) | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 5 | 6
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 4
Colitis ischaemic (Gastrointestinal disorders) | 5 | 1
Gastric ulcer (Gastrointestinal disorders) | 5 | 1
Ileus (Gastrointestinal disorders) | 4 | 5
Large intestine polyp (Gastrointestinal disorders) | 4 | 5
Pancreatitis acute (Gastrointestinal disorders) | 4 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 4 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 7
Abdominal hernia (Gastrointestinal disorders) | 3 | 6
Melaena (Gastrointestinal disorders) | 3 | 4
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 3 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 3
Haemorrhoids (Gastrointestinal disorders) | 3 | 2
Ascites (Gastrointestinal disorders) | 3 | 1
Diverticulum (Gastrointestinal disorders) | 3 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 3 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 3 | 1
Haematemesis (Gastrointestinal disorders) | 3 | 0
Hiatus hernia (Gastrointestinal disorders) | 2 | 5
Obstructive pancreatitis (Gastrointestinal disorders) | 2 | 4
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 3
Duodenal ulcer (Gastrointestinal disorders) | 2 | 2
Anal fistula (Gastrointestinal disorders) | 2 | 1
Large intestine perforation (Gastrointestinal disorders) | 2 | 1
Peptic ulcer (Gastrointestinal disorders) | 2 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 2 | 0
Gastritis erosive (Gastrointestinal disorders) | 2 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 2 | 0
Retroperitoneal fibrosis (Gastrointestinal disorders) | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 10
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 3
Haematochezia (Gastrointestinal disorders) | 1 | 2
Diverticular perforation (Gastrointestinal disorders) | 1 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Peritoneal disorder (Gastrointestinal disorders) | 1 | 1
Appendix disorder (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Duodenogastric reflux (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 | 0
Proctitis ulcerative (Gastrointestinal disorders) | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 2
Food poisoning (Gastrointestinal disorders) | 0 | 2
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 2
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Duodenitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Mesenteric arterial occlusion (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal pain (Gastrointestinal disorders) | 0 | 1
Pancreatic mass (Gastrointestinal disorders) | 0 | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 81 | 73
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 11
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 16 | 7
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 11 | 5
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 10 | 12
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 10 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 3
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 4
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 4
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Mandibular mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatic fever (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 5
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 33 | 34
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 19 | 18
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 13
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 14 | 22
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 16 | 15
Subdural haematoma (Injury, poisoning and procedural complications) | 9 | 5
Hip fracture (Injury, poisoning and procedural complications) | 8 | 8
Incisional hernia (Injury, poisoning and procedural complications) | 6 | 3
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 5 | 3
Rib fracture (Injury, poisoning and procedural complications) | 5 | 3
Head injury (Injury, poisoning and procedural complications) | 5 | 2
Femur fracture (Injury, poisoning and procedural complications) | 4 | 10
Ankle fracture (Injury, poisoning and procedural complications) | 4 | 5
Tendon rupture (Injury, poisoning and procedural complications) | 4 | 4
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 4 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 4
Laceration (Injury, poisoning and procedural complications) | 3 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 3 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 3
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 2
Ligament injury (Injury, poisoning and procedural complications) | 2 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 2 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 2 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 2 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 2 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 2
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0
Bone fragmentation (Injury, poisoning and procedural complications) | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of sternum (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 1 | 0
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 | 0
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 | 0
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 2
Brain contusion (Injury, poisoning and procedural complications) | 0 | 2
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2
Stomal hernia (Injury, poisoning and procedural complications) | 0 | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Axillary nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Oesophageal injury (Injury, poisoning and procedural complications) | 0 | 1
Poisoning deliberate (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Radiation injury (Injury, poisoning and procedural complications) | 0 | 1
Sciatic nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Traumatic renal injury (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1
Urethral injury (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Chest pain (General disorders) | 66 | 66
Non-cardiac chest pain (General disorders) | 49 | 52
Asthenia (General disorders) | 6 | 8
Malaise (General disorders) | 5 | 3
Pyrexia (General disorders) | 4 | 5
Oedema peripheral (General disorders) | 3 | 2
Multiple organ dysfunction syndrome (General disorders) | 2 | 1
General physical health deterioration (General disorders) | 2 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 7
Chest discomfort (General disorders) | 1 | 4
Fatigue (General disorders) | 1 | 2
Cyst (General disorders) | 1 | 1
Impaired healing (General disorders) | 1 | 1
Adverse drug reaction (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Complication associated with device (General disorders) | 1 | 0
Drowning (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Swelling (General disorders) | 1 | 0
Ulcer (General disorders) | 1 | 0
Ulcer haemorrhage (General disorders) | 1 | 0
Vascular stent restenosis (General disorders) | 1 | 0
Exercise tolerance decreased (General disorders) | 0 | 3
Incarcerated hernia (General disorders) | 0 | 2
Polyp (General disorders) | 0 | 2
Catheter site haemorrhage (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pelvic mass (General disorders) | 0 | 1
Suprapubic pain (General disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 47 | 34
Nephrolithiasis (Renal and urinary disorders) | 13 | 12
Renal failure (Renal and urinary disorders) | 11 | 6
Haematuria (Renal and urinary disorders) | 8 | 4
Ureterolithiasis (Renal and urinary disorders) | 6 | 7
Chronic kidney disease (Renal and urinary disorders) | 6 | 4
Urinary retention (Renal and urinary disorders) | 5 | 4
Renal impairment (Renal and urinary disorders) | 5 | 1
Renal cyst (Renal and urinary disorders) | 4 | 0
Urethral stenosis (Renal and urinary disorders) | 3 | 2
Urinary tract obstruction (Renal and urinary disorders) | 3 | 1
Calculus urinary (Renal and urinary disorders) | 2 | 3
Renal colic (Renal and urinary disorders) | 2 | 3
End stage renal disease (Renal and urinary disorders) | 2 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 2 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 2
Stress urinary incontinence (Renal and urinary disorders) | 1 | 2
Bladder neck obstruction (Renal and urinary disorders) | 1 | 1
Nephropathy (Renal and urinary disorders) | 1 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 1
Bladder stenosis (Renal and urinary disorders) | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 0
Renal artery fibromuscular dysplasia (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal injury (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Ureteric dilatation (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 0
Urethral meatus stenosis (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 4
Urinary incontinence (Renal and urinary disorders) | 0 | 4
Acute prerenal failure (Renal and urinary disorders) | 0 | 2
Bladder dysfunction (Renal and urinary disorders) | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Stag horn calculus (Renal and urinary disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1
Syncope (Nervous system disorders) | 28 | 31
Dizziness (Nervous system disorders) | 11 | 10
Transient ischaemic attack (Nervous system disorders) | 8 | 3
Encephalopathy (Nervous system disorders) | 7 | 2
Presyncope (Nervous system disorders) | 6 | 6
Cerebrovascular accident (Nervous system disorders) | 3 | 5
Headache (Nervous system disorders) | 3 | 4
Seizure (Nervous system disorders) | 3 | 4
Metabolic encephalopathy (Nervous system disorders) | 2 | 3
Carpal tunnel syndrome (Nervous system disorders) | 2 | 1
Cervical radiculopathy (Nervous system disorders) | 2 | 1
Ataxia (Nervous system disorders) | 2 | 0
Dementia (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 2 | 0
Intracranial aneurysm (Nervous system disorders) | 2 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 3
Neuralgia (Nervous system disorders) | 1 | 2
Aphasia (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 1
Facial paralysis (Nervous system disorders) | 1 | 1
Hydrocephalus (Nervous system disorders) | 1 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Transient global amnesia (Nervous system disorders) | 1 | 1
Unresponsive to stimuli (Nervous system disorders) | 1 | 1
Brain injury (Nervous system disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Dural arteriovenous fistula (Nervous system disorders) | 1 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0
Intracranial mass (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0
Neurodegenerative disorder (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 1 | 0
Pseudoradicular syndrome (Nervous system disorders) | 1 | 0
Quadriplegia (Nervous system disorders) | 1 | 0
Radicular syndrome (Nervous system disorders) | 1 | 0
Sensory ganglionitis (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Trigeminal nerve disorder (Nervous system disorders) | 1 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 5
Cerebral haemorrhage (Nervous system disorders) | 0 | 2
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 2
Loss of consciousness (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 0 | 2
Acute disseminated encephalomyelitis (Nervous system disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1
Carotid artery disease (Nervous system disorders) | 0 | 1
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 | 1
Spinal cord herniation (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Vascular dementia (Nervous system disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 16 | 11
Hypoglycaemia (Metabolism and nutrition disorders) | 15 | 14
Diabetes mellitus (Metabolism and nutrition disorders) | 11 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 8
Obesity (Metabolism and nutrition disorders) | 9 | 5
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 2 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Shock hypoglycaemic (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperosmolar state (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 15 | 11
Hypertension (Vascular disorders) | 12 | 16
Hypotension (Vascular disorders) | 9 | 11
Deep vein thrombosis (Vascular disorders) | 5 | 8
Aortic stenosis (Vascular disorders) | 4 | 10
Orthostatic hypotension (Vascular disorders) | 4 | 5
Aortic aneurysm (Vascular disorders) | 3 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 3
Hypovolaemic shock (Vascular disorders) | 2 | 1
Accelerated hypertension (Vascular disorders) | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 2 | 0
Shock haemorrhagic (Vascular disorders) | 2 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 3
Peripheral artery occlusion (Vascular disorders) | 1 | 2
Aortic aneurysm rupture (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 1 | 1
Hypertensive emergency (Vascular disorders) | 1 | 1
Intermittent claudication (Vascular disorders) | 1 | 1
Shock (Vascular disorders) | 1 | 1
Angiodysplasia (Vascular disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Embolism arterial (Vascular disorders) | 1 | 0
Extravasation blood (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
Renovascular hypertension (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Leriche syndrome (Vascular disorders) | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 15 | 18
Cholecystitis acute (Hepatobiliary disorders) | 15 | 7
Cholecystitis (Hepatobiliary disorders) | 9 | 7
Cholangitis (Hepatobiliary disorders) | 4 | 1
Bile duct stone (Hepatobiliary disorders) | 3 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 3 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 1
Alcoholic liver disease (Hepatobiliary disorders) | 1 | 0
Cryptogenic cirrhosis (Hepatobiliary disorders) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 2
Gallbladder enlargement (Hepatobiliary disorders) | 0 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 2
Biliary colic (Hepatobiliary disorders) | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 22 | 20
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 3
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Splenic infarction (Blood and lymphatic system disorders) | 0 | 2
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 18 | 11
Prostatitis (Reproductive system and breast disorders) | 6 | 3
Prostatomegaly (Reproductive system and breast disorders) | 2 | 2
Adnexa uteri mass (Reproductive system and breast disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 1 | 0
Peyronie's disease (Reproductive system and breast disorders) | 1 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 2
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Endometrial hypoplasia (Reproductive system and breast disorders) | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1
Seminal vesicular cyst (Reproductive system and breast disorders) | 0 | 1
Testicular cyst (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Delirium (Psychiatric disorders) | 5 | 2
Suicide attempt (Psychiatric disorders) | 3 | 1
Mental status changes (Psychiatric disorders) | 2 | 3
Depression (Psychiatric disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 2 | 0
Panic attack (Psychiatric disorders) | 2 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 3
Completed suicide (Psychiatric disorders) | 1 | 2
Suicidal ideation (Psychiatric disorders) | 1 | 2
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Aggression (Psychiatric disorders) | 1 | 0
Agitated depression (Psychiatric disorders) | 1 | 0
Delirium tremens (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Schizoaffective disorder (Psychiatric disorders) | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 | 3
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 2
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 2 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Granuloma annulare (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 3 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 2 | 1
Lung lobectomy (Surgical and medical procedures) | 1 | 1
Aortic valve replacement (Surgical and medical procedures) | 1 | 0
Artificial urinary sphincter implant (Surgical and medical procedures) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0
Polypectomy (Surgical and medical procedures) | 1 | 0
Rotator cuff repair (Surgical and medical procedures) | 1 | 0
Shoulder operation (Surgical and medical procedures) | 1 | 0
Stem cell transplant (Surgical and medical procedures) | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0
Cardiac ablation (Surgical and medical procedures) | 0 | 2
Spinal operation (Surgical and medical procedures) | 0 | 2
Endotracheal intubation (Surgical and medical procedures) | 0 | 1
Gastric bypass (Surgical and medical procedures) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Large intestinal polypectomy (Surgical and medical procedures) | 0 | 1
Transurethral bladder resection (Surgical and medical procedures) | 0 | 1
Troponin increased (Investigations) | 2 | 3
Arteriogram coronary (Investigations) | 2 | 1
Ejection fraction decreased (Investigations) | 2 | 1
Blood pressure increased (Investigations) | 1 | 2
Blood glucose increased (Investigations) | 1 | 1
Weight decreased (Investigations) | 1 | 1
Biopsy pleura (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Influenza A virus test positive (Investigations) | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 2
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1
Blood pressure difference of extremities (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Ejection fraction abnormal (Investigations) | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Influenza virus test positive (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Cataract (Eye disorders) | 4 | 5
Retinal detachment (Eye disorders) | 3 | 0
Eyelid ptosis (Eye disorders) | 1 | 1
Retinal haemorrhage (Eye disorders) | 1 | 1
Diplopia (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 2
Chalazion (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 5 | 8
Vertigo positional (Ear and labyrinth disorders) | 2 | 5
Vestibular disorder (Ear and labyrinth disorders) | 0 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 1
Inner ear disorder (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Device malfunction (Product Issues) | 2 | 2
Device breakage (Product Issues) | 1 | 2
Device dislocation (Product Issues) | 1 | 2
Device failure (Product Issues) | 1 | 2
Device occlusion (Product Issues) | 0 | 1
Thyroid mass (Endocrine disorders) | 2 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 4
Addison's disease (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 2
Hypersensitivity (Immune system disorders) | 1 | 1
Allergy to arthropod sting (Immune system disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 2 | 0
Pancreas divisum (Congenital, familial and genetic disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMR101 (N=4089) | Placebo (N=4090)
Anaemia (Blood and lymphatic system disorders) | 178 | 224
Cataract (Eye disorders) | 230 | 205
Diarrhoea (Gastrointestinal disorders) | 363 | 450
Constipation (Gastrointestinal disorders) | 216 | 142
Oedema peripheral (General disorders) | 264 | 201
Fatigue (General disorders) | 227 | 195
Chest pain (General disorders) | 226 | 240
Nasopharyngitis (Infections and infestations) | 314 | 300
Upper respiratory tract infection (Infections and infestations) | 311 | 315
Bronchitis (Infections and infestations) | 295 | 292
Influenza (Infections and infestations) | 261 | 267
Urinary tract infection (Infections and infestations) | 240 | 246
Back pain (Musculoskeletal and connective tissue disorders) | 322 | 303
Arthralgia (Musculoskeletal and connective tissue disorders) | 309 | 306
Pain in extremity (Musculoskeletal and connective tissue disorders) | 232 | 239
Dizziness (Nervous system disorders) | 227 | 238
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 243 | 233
Cough (Respiratory, thoracic and mediastinal disorders) | 241 | 241
Hypertension (Vascular disorders) | 312 | 333

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT01492361/Prot_SAP_000.pdf